CLINICAL TRIAL: NCT02898051
Title: Anti Xa Activity in Cancer Patients Receiving Low-molecular-weight Heparin for Venous Thromboembolism
Acronym: aXa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P100127; PHRC10_02-54 (Other Grant/Funding Number: French Ministry of health); 2011-000154-36 (EudraCT Number)
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms; Venous Thromboembolism
Keywords: heparin low-molecular-weight;pharmacokinetics
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen Description
  The total volume of blood collected for the study will be 44 mL for cancer patients and non cancer patients for the measurement of the following parameters:
  * anti-Xa activity;
  * heparanase;
  * platelet factor 4;
  * tissue factor;
  * tissue factor pathway inhibitor (TFPI);
  * P-selectin.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Venous Thromboembolism and cancer: Patients hospitalized for Venous Thromboembolism and having a cancer. Inclusion (as soon as the diagnosis of venous thromboembolism is confirmed). One tube of blood taken before the start of treatment (at the time of another blood sample) for determination of heparanase. After the start of treatment: three tubes of blood drawn for determination of anti-Xa activity.
  Assays will be centrally performed, blinded from the clinical data and from the group knowledge of the group patient.
- Venous Thromboembolism and non cancer: Patients hospitalized for Venous Thromboembolism and not having a cancer. Inclusion (as soon as the diagnosis of venous thromboembolism is confirmed). One tube of blood taken before the start of treatment (at the time of another blood sample) for determination of heparanase. After the start of treatment: 3 tubes of blood drawn for determination of anti-Xa activity.
  Assays will be centrally performed, blinded from the clinical data and from the group knowledge of the group patient.

SUMMARY:
Low molecular weight heparins (LMWH) are the reference molecule for the long term treatment of venous thromboembolism (VTE) in cancer patients but remains, however, associated with a high risk of recurrent thromboembolism. The high rate of recurrence may result from alterations in the pharmacokinetics of LMWH. The primary purpose of the study is to compare the pharmacokinetics of anti-Xa activity in patients with cancer and patients without cancer treated with curative dose of low molecular weight heparins (LMWH) for venous thromboembolism (VTE). The secondary purposes are 1/ to study the correlation between anti-Xa LMWH and concentration of plasma heparanase and 2/ to evaluate the predictive nature of the anti-Xa activity on the occurrence of thromboembolic recurrence in cancer patients treated with LMWH for VTE.

DETAILED DESCRIPTION:
Purpose of the study:

The primary purpose of the study is to compare the pharmacokinetics of anti-Xa activity in patients with cancer and patients without cancer treated with curative dose of low molecular weight heparins (LMWH) for venous thromboembolism (VTE).

The secondary purposes are 1/ to study the correlation between anti-Xa LMWH and concentration of plasma heparanase and 2/ to evaluate the predictive nature of the anti-Xa activity on the occurrence of thromboembolic recurrence in cancer patients treated with LMWH for VTE.

Study design:

Multicentre cohort study of patients hospitalized with VTE:

1. Observational case-control study to compare the pharmacodynamics of anti-Xa activity between patients cancer patients (n = 50) and non-cancer patients (n = 50) matched (1-1) for age, renal function and LMWH
2. A prospective cohort study including 320 cancer patients with a 6 months follow-up.

Study hypothesis:

Venous thrombosis and pulmonary embolism are a common complication of cancer. They complicate up to 10% of cancers and are the cause of fatality, morbidity and significant impaired quality of life. The treatment of these diseases is difficult in this context. Low molecular weight heparins (LMWH) are the reference molecule for the long term treatment of venous thromboembolism (VTE) in cancer patients. Outside this context, their pharmacological properties allow to administer a fixed dose without measuring anti-Xa activity. In the presence of cancer, their use remains, however, associated with a high risk of recurrent thromboembolism up to 9% after 6 months of treatment.

This high rate of recurrence may result from alterations in the pharmacokinetics of LMWH in the presence of a cancer. The synthesis of heparanase by tumor cells might cause a decrease in anti-Xa activity of LMWH and reduce their effectiveness. If this hypothesis is verified, it could result in a change in the management of thrombosis in cancer patients and lead to a dose adjustment of LMWH through the measurement of anti-Xa activity, which may allow reduce the incidence of thromboembolic relapses during treatment.

Enrollment (Target or Actual Number of Subjects):

1. Pharmacokinetics study In a preliminary unpublished study of 37 cancer and non-cancer subjects with the highest concentration of anti-Xa activity was measured. Included 100 subjects (50 cancer patients and 50 non-cancer) would detect a maximum level difference of anti-Xa activity in plasma of 0.20 between cancer patients and cancer-with a power of 90% and a risk of the first kind 5%.

   A difference of 0.20 seems relevant from these preliminary data (median 0.46 vs 0.65), and returns to show that a cancer patient has over 70% chance of having a maximum concentration of anti-Xa activity below that of a free cancer patient (nonparametric Wilcoxon test).
2. Cohort study (cancer patients) The risk of recurrent thromboembolism was estimated between 5 and 10% in cancer patients. By including 200 subjects, around twenty events would be observed and corresponds to a reasonable number of subjects can be recruited over 18 months (50 would already enroll in the pharmacodynamic study). The event rate will be assessed on the first 100 patients that will have been followed for 6 months, if event rate is lower than expected, the number of participants will be reassessed.

After over 2 years of inclusion, the event rate is lower than expected (7%). The number of subjects required was therefore reassessed. To reach the number of 20 events necessary to our analysis, a total of 320 cancer subjects must therefore be included.

Target Follow-Up, duration :

Study duration: 5 years and 6 months (inclusion: 5 years follow-up: 6 months). Duration of participation: 3 a 10 days for non-cancer patients, 6 months for cancer patient.

Performance of the study:

1. Pharmacokinetics study Inclusion (as soon as the diagnosis is confirmed VTE): 1 tube of blood taken before the start of treatment (at the time of another blood sample) for determination of heparanase. After the start of treatment: 3 tubes of blood drawn for determination of anti-Xa activity.

   Assays will be centrally performed, blinded from the clinical data and from the group knowledge of the group patient.
2. Prospective cohort study of cancer patients Followed for 6 months with consultation at 1, 3, and 6 months (normal monitoring).

Follow-up visits: Collection of clinical data (recurrent thromboembolism, hemorrhage, death, tumor progression, cancer treatment since last visit, interruption of treatment with LMWH, thrombocytopenia, anemia), and removal of 1 tube of blood (at the time of a another sample) for determination of anti-Xa activity.

Thromboembolic recurrences will be validated centrally by an independent committee.

Prospects:

Reduce the incidence of thromboembolic recurrence in cancer patients treated with LMWH for VTE by adapting the dose of LMWH with anti-Xa activity in this population if the hypothesis is verified.

ELIGIBILITY:
Inclusion Criteria:

Case:

* Being affiliated to a social security scheme
* Having an active solid or hematological cancer (myeloma or lymphoma), histologically or cytologically confirmed, for which the active state will be defined by the existence of a tumoral active disease or an incomplete tumoral resection or the persistence of high tumor markers after complete resection of the tumor.
* The venous thromboembolism disease has to be:
* A deep vein thrombosis of lower extremity (proximal or distal) confirmed by the lack of compressibility of a venous segment under the ultrasound probe or the presence of a venous gap in CT venography or phlebography;
* or a thrombosis of the vena cava or the iliac vein confirmed by an abdominal CT scan with contrast or a venous ultrasound or an ilio-cavography;
* or a pulmonary embolism confirmed according to the guidelines of the European Society of Cardiology : through a gap in a pulmonary artery, at least segmental or multiple gaps sub-segmental on spiral CT angiography of the pulmonary arteries or by a high appearance probability on a lung radionuclide imaging, or by clinical symptoms of pulmonary embolism accompanying symptomatic proximal vein thrombosis confirmed by a venous ultrasound or by an unexplained echocardiography acute pulmonary heart in presence of a high clinical probability and for patients who are unfit for transport and with cardiogenic shock
* The venous thromboembolism disease can be asymptomatic or incidentally discovered but is confirmed objectively.
* No cons-indication to low molecular weight heparin treatment at therapeutic dose.
* Prescription in the last 72 hours of a low molecular weight heparin treatment or fondaparinux at therapeutic dose.

Control:

* Being affiliated to a social security scheme.
* Being free from malignant tumor pathology detectable at the time of inclusion.
* Being afflicted with venous thromboembolism defined by the same criteria of cancer subjects.
* The venous thromboembolism disease can be asymptomatic or incidentally discovered but is confirmed objectively.
* No cons-indication to low molecular weight heparin treatment at therapeutic dose.
* Prescription in the last 72 hours of a low molecular weight heparin treatment or fondaparinux at therapeutic dose.

Exclusion Criteria:

Case:

* Visceral vein thrombosis of the upper limb or venous thrombosis of the superior vena cava system because their scalability under treatment, including the risk of embolic recurrence is less known that pulmonary embolism and thrombosis of the lower limbs and their diagnostic modalities are less formalized.
* Tumor disease not confirmed histologically or cytologically.
* Follow-up after complete tumor resection without elevated tumor markers.
* Cons-indication to low molecular weight heparin treatment at therapeutic dose.
* Initial treatment with another anticoagulant molecule than LMWH or fondaparinux (thrombin inhibitor, direct factor Xa inhibitors)
* Severe renal impairment defined by a creatinine clearance below than 30 ml / min at baseline.
* Known pregnancy or lack of effective contraception for women of childbearing age or breastfeeding.
* Patient previously included in the study.
* Impossible follow-up.
* Life expectancy less than 6 months.
* Patient whose weight is greater than 100 Kg.

Control:

* Not yet confirmed suspected malignant tumor pathology associated with the venous thromboembolism disease.
* Active cancer in the last 2 years.
* Cons-indication to low molecular weight heparin treatment at therapeutic dose.
* Initial treatment with another anticoagulant molecule than LMWH or fondaparinux (thrombin inhibitor, direct factor Xa inhibitors)
* Severe renal impairment defined by a creatinine clearance below than 30 ml / min at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in tertiary care hospitals participating to the study and treated with curative dose of low molecular weight heparins (LMWH) for venous thromboembolism (VTE).
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
anti-Xa activity | 10 days
  The measurement of anti-Xa activity will be performed four times during the initial treatment for each patient (or during the first 5 to 10 days of treatment) and will establish pharmacokinetic modeling (population type approach, nonlinear model mixed-effect) of the low molecular weight heparin therapy in subjects with cancer or not. In order to obtain a curve of relevant anti-Xa activity.

SECONDARY OUTCOMES:
hemorrhage | 6 months
  Major hemorrhage:
  * hemorrhage at the origin of death;
  * symptomatic hemorrhage in a major organ such as intracranial hemorrhage, intra spinal, intraocular, retro peritoneal, intra-articular, pericardial and muscle bleeding causing a compartment syndrome
  * symptomatic hemorrhage causing a fall in hemoglobin of at least 2 g / dL or leading to a transfusion of at least two blood units.
  Other hemorrhage will be considered as non-major.
all cause mortality | 6 months
  Cause and date of death.
  The death will be classified as follows:
  * related to cancer;
  * secondary to bleeding;
  * secondary to a confirmed pulmonary embolism;
  * other cause;
  * unexplained sudden death that can be attributed to pulmonary embolism.
thromboembolic recurrences | 6 months
  All thromboembolic events diagnosed during the follow-up period will be considered in the analysis, whether symptomatic or discovered incidentally on radiographic examination for another reason, evaluation of tumor progression in particular. The recurrence of venous thrombosis should be confirmed objectively by the presence of a non-compressible venous segment in an initially compressible area or by the appearance of a new gap in the CT venography.
  The recurrence of pulmonary embolism must be confirmed by the appearance of a gap in a normal artery on the initial scanner or the more proximal extension of thrombosis on the 2nd scanner or the appearance of a segmental perfusion defect without abnormality of ventilation in an initially normal part on the initial scintigraphy or the initial scan.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Meyer, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (8):
- France (8):
  - Hôpital d'instruction des armees Desgenettes, Lyon, Auvergne-Rhône-Alpes
  - CHU de Saint-Etienne Hôpital Nord, Saint-Priest-en-Jarez, Auvergne-Rhône-Alpes
  - CHU de Dijon, Dijon, Bourgogne-Franche-Comté
  - Hôpital La Cavale Blanche, Brest, Brittany Region
  - CHU Amiens - Hôpital Sud, Amiens, Picardie
  - Hôpital Louis Mourier, Colombes, Île-de-France Region
  - Hôpital Saint-Louis, Paris, Île-de-France Region
  - Hôpital Europeen Georges Pompidou, Paris, Île-de-France Region

REFERENCES:
- [Background] Chew HK, Wun T, Harvey D, Zhou H, White RH. Incidence of venous thromboembolism and its effect on survival among patients with common cancers. Arch Intern Med. 2006 Feb 27;166(4):458-64. doi: 10.1001/archinte.166.4.458. PMID 16505267
- [Background] Khorana AA, Streiff MB, Farge D, Mandala M, Debourdeau P, Cajfinger F, Marty M, Falanga A, Lyman GH. Venous thromboembolism prophylaxis and treatment in cancer: a consensus statement of major guidelines panels and call to action. J Clin Oncol. 2009 Oct 10;27(29):4919-26. doi: 10.1200/JCO.2009.22.3214. Epub 2009 Aug 31. PMID 19720907
- [Background] Kearon C, Kahn SR, Agnelli G, Goldhaber S, Raskob GE, Comerota AJ. Antithrombotic therapy for venous thromboembolic disease: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):454S-545S. doi: 10.1378/chest.08-0658. PMID 18574272
- [Background] Lee AY, Levine MN, Baker RI, Bowden C, Kakkar AK, Prins M, Rickles FR, Julian JA, Haley S, Kovacs MJ, Gent M; Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer (CLOT) Investigators. Low-molecular-weight heparin versus a coumarin for the prevention of recurrent venous thromboembolism in patients with cancer. N Engl J Med. 2003 Jul 10;349(2):146-53. doi: 10.1056/NEJMoa025313. PMID 12853587
- [Background] Katz BZ, Muhl L, Zwang E, Ilan N, Herishanu Y, Deutsch V, Naparstek E, Vlodavsky I, Preissner KT. Heparanase modulates heparinoids anticoagulant activities via non-enzymatic mechanisms. Thromb Haemost. 2007 Dec;98(6):1193-9. PMID 18064313